CLINICAL TRIAL: NCT02298933
Title: Complement Inhibition Using Eculizumab to Overcome Platelet Transfusion Refractoriness in Patients With Severe Thrombocytopenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150015; 15-H-0015
Record Dates: First submitted 2014-11-21; First posted 2014-11-24 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-01-18

CONDITIONS: Thrombocytopenia; Alloimmune Platelet Refractoriness
Keywords: Complement Inhibition; Platelet Refractoriness; Eculizumab
MeSH Terms: conditions — Thrombocytopenia | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eculizumab (Experimental): 1200 mg IV infusion over 30-40 min
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — 300 mg single-use vials

SUMMARY:
Background:

- Platelets are tiny cells in the blood that help stop bleeding. Thrombocytopenia happens when people do not have enough normal platelets. Getting a transfusion of another person s platelets can help stop too much bleeding. But because these cells are from other people, the body may reject them,putting them at risk for serious bleeding complications. This conditions is called alloimmune platelet refractoriness . There are evidence that in many patients, platelet counts fail to increase after a platelet transfusion because the transfused platelets are destroyed by the body s defence soldier, called complement . Researchers want to see if a drug, that inhibits complement, can help increase platelet levels and reduce bleeding

Objectives:

- To see if eculizumab increases platelet levels more after a transfusion. To see if it reduces the chance of bleeding too much.

Eligibility:

- Adults 18-75 years old who have thrombocytopenia and alloimmune platelet refractoriness.

Design:

* Participants will be screened with medical history, physical exam, and blood tests.
* Participants will have the procedures listed below. They can have them while they are in the hospital. Or they can go to the outpatient clinic for them. Each visit may take up to 3 hours.
* Participants will get a meningitis vaccine if needed. Then they will get the study drug as an infusion.
* Participants will have a platelet transfusion. Their blood will be drawn every 24 hours until the platelet count is less than 10,000 per 1 microliter of blood.
* They will take antibiotics for 14 days.
* Participants will have a checkup and blood drawn twice a week for 2 weeks. They will get more transfusions if needed.

DETAILED DESCRIPTION:
Platelet transfusion can be a life-saving procedure in preventing or treating serious bleeding in patients who have low and/or dysfunctional platelets. Treatment of blood cancer and other blood diseases as well as bone marrow transplantation is not possible without platelet transfusion support. Unfortunately, 20-60% of chronically transfused patients will stop responding to these transfusions putting them at risk for serious bleeding complications. Data support the concept that in many patients, platelet counts fail to increase after a platelet transfusion because the transfused platelets are destroyed by the body s complement. In order to overcome this problem, we will inhibit complement activity with the medication eculizumab that specifically binds and suppresses complement. We hypothesize that when we treat patients who have platelet refractoriness with eculizumab, the platelet counts will increase to higher numbers after platelet transfusions, decreasing the risk of bleeding complications associated with having a low platelet count.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Ages 18-75 years inclusive.
* Ability to comprehend the investigational nature of the study and provide informed consent.
* Thrombocytopenia (due to congenital causes, bone marrow failure, hematologic malignancies, and treatment related), defined as <10k/uL without bleeding or <30K/uL with evidence of life threatening bleeding (intracranial hemorrhage, GI bleeding, pulmonary hemorrhage, uncontrolled epistaxis, hematuria).
* Diagnosed with immune platelet refractoriness, characterized by all of the following:

  * Lack of adequate post-transfusion platelet count increment, defined by, CCI <7500/ul at 10-60 min, and CCI <5000/ul at 18-24 hrs (in those who had a CCI at 10-60 min greater than or equal to 5000/microl)after at least 2 consecutive transfusions.
  * Presence of anti-HLA class A and/or B antibody.

EXCLUSION CRITERIA:

* Active meningococcal infection.
* Severe psychiatric illness. Mental deficiency sufficiently severe as to make making informed consent impossible.
* Positive pregnancy test for women of childbearing age within 1 week.
* HIV positive test within 3 months
* Paroxysmal Nocturnal Hemoglobinuria (PNH) disease with evidence of intravascular hemolysis.
* Presence ITP/autoimmune thrombocytopenia
* Immune platelet refractoriness responsive to treatment with IVIG

RE-ENROLLMENT CRITERIA:

* Meet response criteria to the initial treatment or second treatment
* Meets all initial inclusion/exclusion criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11-21; Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Aue, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Vo P, Purev E, West KA, McDuffee E, Worthy T, Cook L, Hawks G, Wells B, Shalabi R, Flegel WA, Adams SD, Reger R, Aue G, Tian X, Childs R. A pilot trial of complement inhibition using eculizumab to overcome platelet transfusion refractoriness in human leukocyte antigen allo-immunized patients. Br J Haematol. 2020 May;189(3):551-558. doi: 10.1111/bjh.16385. Epub 2020 Feb 21. PMID 32086819
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-H-0015.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Eculizumab: Eculizumab 1200 mg IV infusion is given over 30-40 min
Period: Overall Study
Arm/Group | Eculizumab
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eculizumab
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Sustained Platelet Transfusion Responsiveness
Description: To evaluate the safety and efficacy of eculizumab to increase the platelet increment, defined as Corrected Count Increment (CCI) >7500/μL at 10-60 min together with CCI>5000/μL at 18-24 hrs post transfusion in patients with platelet refractoriness following treatment with eculizumab and platelet transfusion.
Time Frame: 24 hours
Population: All patients were given Eculizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 10
Participants | 4

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Eculizumab
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 6/10
Other Adverse Events (participants affected / at risk) | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=10)
Pericardial effusion (Cardiac disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Infection (Infections and infestations) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Dyspnoea (Cardiac disorders) | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1
Eye disorder (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Decreased appetite (General disorders) | 1
Pyrexia (General disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Tremor (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT02298933/Prot_SAP_000.pdf